CLINICAL TRIAL: NCT05070273
Title: Safety and Feasibility of St. Mark's Electrode for the Hypoglossal Nerve and Cortico-lingual Pathway Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NMSC-03-21
Record Dates: First submitted 2021-09-23; First posted 2021-10-07 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
Keywords: hypoglossal nerve

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoglossal nerve conduction study. (Experimental)
  Interventions: Diagnostic Test: Hypoglossal nerve conduction study; Diagnostic Test: Transcranial magnetic stimulation of hypoglossal nerve

INTERVENTIONS:
Diagnostic Test: Hypoglossal nerve conduction study — NCS of nervus hypoglossus (evaluation of M-response parameters) was carried out using a 4-channel electromyographic machine. The stimulation will be carried out from three points:
  1. angle of the lower jaw (proximal point),
  2. the area of the carotid triangle (distal point),
  3. directly from the electrode of St. Mark when it is localized on the muscles of the tongue.
  The initial stimulation parameters: strength of an electric current 20 mA, stimulus duration 0.2 ms, and frequency 1 Hz. To achieve supramaximal stimulation, the stimulation strength will be increased with a step of 1-2 mA to a maximum of 35 mA, the duration of the stimulus will be increased to 0.3 ms.
Diagnostic Test: Transcranial magnetic stimulation of hypoglossal nerve — TMS will be carried out using a Magstim 200 magnetic stimulator connected with a BiStim module (Magstim Co. Ltd., Whitland, Wales, UK). The generated magnetic pulses will be delivered by the coil 65 mm in diameter tangentially located relative to the scalp in the F7 projection - T3 and F8-T4 (according to the international scheme "10-20"). The area of cortical stimulation will be localized by supplying single pulses with gradual increase, with a coil displacement with a step of 1 cm, until the contraction of the facial muscles will be obtained, followed by the determination of the MEP threshold value. Analysis of conduction by cortical-lingual pathway will be performed at TMS with magnetic stimulus intensity 20-30% above the MEP threshold.

SUMMARY:
The possibility of registering the M-response and the motor evoked potential (MEP) from the muscles of the tongue by using the St. Mark's electrode will be evaluated. The safety of method will be confirmed. Registered parameters will be compared with other known methods and comparative effectiveness of proposed method will be determined.

The study will involve healthy volunteers without clinical symptoms of hypoglossal nerve and cortico-lingual pathway lesions and without surgical interventions in the tongue .The volunteers will be examined once for the parameters of the amplitude and latency of the M-response and MEP, as well as the difference between these indicators at different sides of the examination during nerve conduction study (NCS) and transcranial magnetic stimulation (TMS) of the hypoglossal nerve and the cortico-lingual pathway.

ELIGIBILITY:
Inclusion criteria:

* Absence of clinical symptoms of impaired hypoglossal nerve and cortico-lingual pathways;
* Absence of history of surgical interventions in the tongue area;
* The subject has read the information sheet and signed the informed consent.

Exclusion Criteria:

* Clinical symptoms of hypoglossal nerve or cortico-lingual pathway (dysarthria, dysphagia (pseudobulbar palsy) lesions, flaccid paralysis of the tongue muscles, atrophy and fasciculations of the tongue muscles);
* Tumors, metastatic lesions and cysts in the region of the brain stem, posterior cranial fossa, base of the skull, in the region of the carotid segment, salivary glands;
* Vascular pathologies in the carotid sinus area: vascular malformations, dissection of the internal carotid artery aneurysm, venous thrombosis;
* Recent dental procedures with one of the following complications: development of an abscess, direct injury to the nerve by medical equipment, development of hematoma;
* History of carotid endarterectomy;
* Motor neuron disease and other neurodegenerative or demyelinating diseases;
* History of cancer and courses of radiation therapy;
* The presence of implantable programmable devices.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Severe adverse reactions and events rate | During the intervention and 1 day after the intervention
  Severe adverse reactions and events will be monitored and registered during procedure of nerve stimulation and on the day of study

SECONDARY OUTCOMES:
Rate of M-wave registration during NCS of hypoglossus nerve using the St. Mark's electrode in healthy volunteers. | During the intervention
  M-wave will be recorded during NCS from three points: A - the angle of the lower jaw (proximal point); B - the area of the carotid triangle (distal point); C - directly from the electrode of St. Mark when it is located on the muscles of the tongue. Stimulation will be carried out with stimuli with a duration of 0.2 ms, a frequency of 1 Hz with a gradual increase in the intensity of the stimulus until supramaximal stimulation will be achieved (maximum up to 35 mA). If necessary, the duration of the stimulus will be increased up to 0.3 ms.
Rate of MEP registration during TMS of cortical-lingual pathway using the St. Mark's electrode in healthy volunteers. | During the intervention
  The generated magnetic pulses will be delivered by the coil 65 mm in diameter tangentially located relative to the scalp in the F7 projection - T3 and F8-T4 (according to the international scheme "10-20"). The area of cortical stimulation will be localized by supplying single pulses with gradual increase, with a coil displacement with a step of 1 cm, until the contraction of the facial muscles will be obtained, followed by the determination of the MEP threshold value. Analysis of conduction by cortical-lingual pathway will be performed at TMS with magnetic stimulus intensity 20-30% above the MEP threshold.

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2 months after completion of the study
Access Criteria: upon the request